CLINICAL TRIAL: NCT05443490
Title: Randomized, Double Blind, Placebo-controlled Clinical Trial to Evaluate the Effect of a Probiotic Mixture in the Treatment of Atopic Dermatitis in Children From 0 to 3 Years Old
Brief Title: Clinical Trial to Evaluate the Effect of a Probiotic Mixture in the Treatment of Atopic Dermatitis in Children
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Bionou Research, S.L. (Network)
Collaborators: Biopolis S.L. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ATOP_PRO.3
Record Dates: First submitted 2022-06-29; First posted 2022-07-05 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic | interventions — maltodextrin

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Double-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Probiotic group (Experimental): Probiotic mixture
  Interventions: Dietary Supplement: Probiotic mixture with three bacterial strains with maltodextrin as a carrier.
- Placebo group (Placebo Comparator): Maltodextrine
  Interventions: Other: Placebo comparator with maltodextrin as a carrier.

INTERVENTIONS:
Dietary Supplement: Probiotic mixture with three bacterial strains with maltodextrin as a carrier. — Sachets containing a probiotic mixture at concentrations equal to or greater than 1x10^9 colony forming unit (CFU) per dose, with maltodextrin as excipient.
  Arms: Probiotic group
Other: Placebo comparator with maltodextrin as a carrier. — Sachets containing maltodextrin
  Arms: Placebo group

SUMMARY:
A prospective case-control multicentric pilot study of 12 weeks duration to evaluate the effect of a probiotic mixture in the treatment of atopic dermatitis in children from 0 to 3 years old, by measuring the severity of the condition using the SCORAD index, as well as the Clinical Global Impression rating scale, the potential decrease in the use of corticosteroids and antihistamines, and the safety of the treatment under study by the number of adverse events related to the product under study.

DETAILED DESCRIPTION:
Atopic dermatitis is a chronic inflammatory disease of the skin, which first symptoms usually develop during childhood, and approximately 50% of cases are diagnosed in the first year of life.

The diagnosis of atopic dermatitis is clinical, because there are no specific microscopic or laboratory changes. One aspect of establishing the diagnosis is the measurement of the severity of the process in these patients. In this regard, one of the best validated methods, more contrasted, more accepted, used and most recommended is the composite scale called index SCORAD (Scoring Atopic Dermatitis). This index consists of a scoring system that takes into account the extent and intensity of five fundamental types of lesions (erythema, edema / papule, exudate / scab, excoriation and lichenification), as well as symptoms (pruritus and loss of sleep) they provoke.

The use of probiotics in the treatment of Atopic Dermatitis has been studied in recent years in a limited number of pilot studies with variable results depending on the probiotic used and the age of the patients included in the study. Recent studies, including a meta-analysis of previous publications, demonstrate a beneficial effect of the use of probiotics in certain circumstances related to age, the type of probiotic used, the dose and combination of probiotics.

In our previous study, the efficacy and safety of the probiotic were demonstrated. The objective of this study is to confirm whether the treatment improves the evolution of the SCORAD index (difference between the values of the first visit and the final one) in children under 4 years of age, comparing the mean of this value in the probiotic group with the control group. For this, a similar methodology will be applied and the same mixture of strains will be used as in the previous study.

Generally speaking, the goals of treatment of atopic dermatitis are to prevent itching, remove exudate, cure the infection, remove the inflammatory lesion, and prevent relapses. To eliminate itching, and the scratching caused by it, recently developed antihistamines are usually used from the acute phase, since the classic ones can present adverse effects on the central nervous system (CNS) that interfere with daily activities. In other hand, in the flare fase or acute exacerbation of atopic dermatitis, topical corticosteroids are used daily, and during the remission phase, weekly regimens can be used.

The main and secondary objectives of this study, aimed to asses the effect of a probiotic mixture in atopic dermatitis are :

PRIMARY OBJECTIVE

Determine if the product under study has an effect on the evolution and treatment of atopic dermatitis, defined as a decrease in the SCORAD index score.

SECONDARY OBJECTIVES

Determine whether the product under study causes a decrease in the use of topical corticosteroids.

Study if the product under study has an effect on the evolution of the Clinical Global Impression (CGI).

Check if the treatment under study reduces the need to use antihistamines. Evaluate the rate of compliance with the treatment during the development of the study.

Study the safety of the treatment under study, defined as the number of adverse events related to the product under study, referred by the patient that occur during the development of the study.

ELIGIBILITY:
Inclusion Criteria:

* Signature of informed consent from the parent / legal guardian of the patient.
* Patients with mild-moderate atopic dermatitis (SCORAD >20).
* Age between 6 months and 3 years old, both inclusive (36 months).
* Patients using topical corticosteroids.
* Diagnosis of atopic dermatitis.

Exclusion Criteria:

* In treatment with phototherapy for atopic dermatitis in the previous 2 months
* In treatment with systemic corticosteroids in the previous month.
* In treatment with immunosuppressants or cytostatics in the previous 2 months.
* Those who have received probiotic treatment in the previous month.
* Those who have been treated with systemic antibiotics in the previous two weeks.
* Patients with axillary or oral temperature > 37.5ºC; or rectal or otic temperature > 38ºC.
* Patients with severe allergic diseases.
* Patients with pathologies related to immunodeficiency or cancer processes.
* Patients with other dermatological pathologies that may make it difficult to assess atopic dermatitis or require the continued use of topical corticosteroids.
* Patients in whom any of the products under study is contraindicated as established in their technical specifications.
* Patients who have participated in drug research studies in the previous 3 months

Ages: 6 Months to 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 150 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2026-10 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in the SCORAD index at 4,8 and 12 weeks | 12 week
  SCORAD index measures the severity of the disease, wich takes into account the extent and intensity of five types of lesions (erythema, edema/papule, exudate/scab, excoriation and lichenification) as well as subjective symptoms (pruritus and loss of sleep).
  Subscales:
  Eczema Spread (A): 0 - 20 Eczema Intensity (B): 0 - 63 Subjective Symptoms (C): 0 - 20
  Total = (A/5) + (Bx7/2) + C Total: 0 - 103 (Higher values represent a worse outcome)

SECONDARY OUTCOMES:
Number of days that each patient requires the administration of topical corticosteroids at 4, 8 and 12 weeks | 12 week
Number of days that each patient requires the administration of topical corticosteroids in disease flares at 4, 8 and 12 weeks | 12 week
Change from baseline in the CGI score at 4,8 and 12 weeks | 12 week
  Clinical Global Impression (CGI) measures the severity of the disease on a 6-point scale, based on the global assessment of the skin lesions.
  Total: 0 - 5 (Higher values represent a worse outcome)
Number of days that each patient requires the administration of antihistamines at 4, 8 and 12 weeks | 12 week
Adherence to the treatment at 4, 8 and 12 weeks | 12 week
  Percentage of treatment intake days

OTHER OUTCOMES:
Number of adverse events from baseline at weeks 4, 8 and 12 | 12 week
  Adverse events referred by the patient's parents that occur during the development of the study

CONTACTS AND LOCATIONS:
Locations (3):
- Hospital del niño Dr. Ovidio Aliaga Uria y Hospital Arco Iris, La Paz, La Paz Department, Bolivia
- Centro de Especialidades Dermatológicas Ac S.A (Dermaláser), San José, Provincia de San José, Costa Rica
- Hospital Universitario del Vinalopó, Elche, Alicante, Spain

IPD SHARING:
Plan to Share IPD: No